CLINICAL TRIAL: NCT06982430
Title: Identification of Predictive Factors for Early Recurrence of Renal Colic Pain After Emergency Department Treatment: A Prospective Study
Brief Title: Early Recurrence of Renal Colic: Predictive Factors
Acronym: ERRC
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Other Study IDs: ERRC
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2022-01

CONDITIONS: Renal Colic; Emergency Department Patient
Keywords: early recurrence, RC pain, emergency department
MeSH Terms: conditions — Renal Colic; Recurrence; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- prospective study of 878 patients
  Interventions: Other: phone call

INTERVENTIONS:
Other: phone call — Included patients were evaluated on day 7 after discharge from the ED through a telephone call.
  This evaluation aimed to identify a recurrence of RC, defined as a NRS score greater than 3 within the 7 days following inclusion and/or a return visit for the same complaint

SUMMARY:
Renal colic (RC) is a common pathology in emergency medicine, with a high risk of recurrence. Early recurrence remains a major concern, affecting up to 30% of patients, with around 84% of these recurrences occurring within two days of the initial episode , despite preventive measures, both pharmacological and non-pharmacological . The recurrence of RC varies significantly between individuals, and systematic evaluation may facilitate personalized treatment . Recurrence is likely influenced by multiple factors, and identifying these could help clinicians develop better preventive strategies.The main aim of our study was to identify factors predictive of early recurrence of RC pain after emergency department (ED) management.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age who were admitted to the ED for acute abdominopelvic pain and whose final diagnosis was RC

Exclusion Criteria:

* patients with documented or suspected pregnancy, and patients without a phone number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: included patients over 18 years of age who were admitted to the ED for acute abdominopelvic pain and whose final diagnosis was RC
Sampling Method: Probability Sample
Enrollment: 878 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
RC recurrence | 7 days
  NRS score greater than 3 within the 7 days following inclusion and/or a return visit for the same complaint

CONTACTS AND LOCATIONS:
Locations (1):
- Nouira Semir, Monastir, Tunisia